CLINICAL TRIAL: NCT06046495
Title: A Phase I Open-label, Multi-dose, Dose Escalation and Dose Expansion Study of the Oral EGFR Inhibitor PLB1004 in Non-Small Cell Lung Cancer
Brief Title: A Study of the Oral EGFR Inhibitor PLB1004 in Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Avistone Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLB1004-I-US01
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PLB1004 (Experimental): PLB1004 given as a mono-therapy in dose escalation and dose expansion phase.
  Interventions: Drug: PLB1004

INTERVENTIONS:
Drug: PLB1004 — PLB1004 will be orally self-administered by the patient as a mono-therapy.

SUMMARY:
This is a Phase I, multicenter, open-label, dose escalation and dose expansion study to assess the safety and pharmacokinetic profile of PLB1004, a mono-anilino-pyrimidine compound, given alone in NSCLC patients with EGFR exon 20 insertion mutations，uncommon mutations, classical mutations (Ex19del and L858R), and drug-resistant mutation (T790M). Patients will be enrolled and dosed according to the most current protocol. This study is made of two Parts. Part 1 includes a dose escalation into 7 cohorts and patient allocation to these cohorts will be via slot allocation. Each cohort has a minimum of 3 and a maximum of 6 patients for a total of 21 - 42 patients. The patient population of the dose escalation phase will include patients with advanced NSCLC harboring EGFR classical mutations or Ex20ins mutations, or uncommon mutations. Part 2 includes an expansion phase and the expansion phase will explore one or more dose levels of PLB1004 in NSCLC patients with EGFR Ex20ins mutations, classical mutations, or uncommon mutations.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document;
2. Male or female adult patients 18 years of age or older;
3. Patients should have recovered from toxicities related to prior anti-tumor therapy;
4. Patients should have recovered from the effects of major surgery;
5. Have a documented EGFR mutation by a local test in tissue or plasma;
6. At least 12 weeks life expectancy;
7. Must have at least one measurable lesion per RECIST v 1.1;
8. Sexually active males and females of childbearing potential must agree to take effective contraceptive measures.

Exclusion Criteria:

1. Received radiotherapy within 14 days before enrollment;
2. Have significant or uncontrolled systemic disease;
3. Have significant or uncontrolled cardiovascular disease;
4. Have had other diagnosed malignant diseases that required treatment within the past 3 years besides NSCLC;
5. Currently have or had a history of interstitial lung disease, drug-induced interstitial lung disease, or radiation pneumonia that requires steroid therapy;
6. Have known hypersensitivity to the similar drugs and excipients of PLB1004;
7. Pregnant or lactating women;
8. Have used other experimental drugs within 2 weeks prior to the first dose of PLB1004;
9. Have any condition or illness that could affect the compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2028-02-09 (Estimated); Study Completion 2028-02-09 (Estimated)

PRIMARY OUTCOMES:
Safety profile of PLB1004 per CTCAE v5.0 | Up to 2 years

SECONDARY OUTCOMES:
To define the DLTs and MTD | Up to 3 years
Area Under the Curve (AUC) of PLB1004 | Approximately 28 days.
Maximum plasma concentration (Cmax) of PLB1004 | Approximately 28 days.
Time to maximum plasma concentration (Tmax) of PLB1004 | Approximately 28 days.
Overall Response Rate (ORR) | Up to 3 years
Progression-Free Survival (PFS) | Up to 3 years
Overall Survival (OS) | Up to 3 years
Disease Control Rate (DCR) | Up to 3 years
Duration of Response (DOR) | Up to 3 years
Change from baseline in corrected QT interval (QTc) using Fridericia formula (QTcF) | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California-Davis, Sacramento, California
  - Research Site, Louisville, Kentucky
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Research Site, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Swedish Health Sciences, Seattle, Washington
  - Research Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No